CLINICAL TRIAL: NCT04322240
Title: Alpha Lipoic Acid and Diabetes Mellitus: Potential Effects on Peripheral Neuropathy and Different Metabolic Parameters
Brief Title: Alpha Lipoic Acid and Diabetes Mellitus: Potential Effects on Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Waleed Ahmed Salaheldeen Hassan, Assistant professor, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Benha22020
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Diabetic Polyneuropathy; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus, Type 2 | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- type 2 DM with peripheral neuropathy (Experimental): Participants will be prescribed 600 mg/day ALA (thiotacid) orally, for 3 months, and will be advised not to discontinue this medication, antidiabetic drugs, or medications used for managing arterial hypertension or dyslipidaemia during the study.
  Interventions: Drug: Alpha lipoic acid

INTERVENTIONS:
Drug: Alpha lipoic acid — Participants will be prescribed 600 mg/day ALA (thiotacid) orally, for 3 months, and will be advised not to discontinue this medication
  Other Names: Thiotacid

SUMMARY:
Patients with type 2 DM who are following will be enrolled into the study. Two visits were scheduled for data collection, physical examination and laboratory testing of the patients: the first prior to initiation of alpha lipoic acid (ALA) administration (baseline visit) and the second at the end of the third month following initiation of ALA (2nd visit).

DETAILED DESCRIPTION:
This prospective, Interventional study will be conducted at Benha university hospital for 3 months. Patients with type 2 DM who are following at the outpatient internal medicine & diabetes Clinics in Benha Univeristy Hospital and are eligible to participate, will be enrolled into the study. Inclusion criteria comprise the following(1) patient's agreement to participate; (2) diabetic peripheral neuropathy diagnosis (3) treatment with alpha lipolic acid (ALA), had to be stable for 3 months during the study.

Two visits were scheduled for data collection, physical examination and laboratory testing of the patients: the first prior to initiation of ALA administration (baseline visit) and the second at the end of the third month following initiation of ALA (2nd visit).

evaluation include:

1. full neurological evaluation including motor, sensory, ankle reflex, Tests for cardiac parasympathetic action
2. nerve conduction study
3. neuromuscular ultrasound
4. HbA1C 5- HDL-C& LDL-C

ELIGIBILITY:
Inclusion Criteria:

* Patient's agreement to participate
* Diabetic peripheral neuropathy

Exclusion Criteria:

* Causes of neuropathy other than diabetes
* Severe renal disease
* Recent treatment for cancer or haematological malignancies;
* Presence of foot ulcers;
* Peripheral arterial disease ;
* Use of agents in the previous 3 months that could interfere with the interpretation of results, such as opiates, vitamin B compounds or antioxidants;
* Pregnancy
* Lactation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
monofilament test of both feet | : through study completion, an average of 3months
  5.07 (10 gram) monofilament will be used to test loss of protective sensation of at 10 sites in each feet at baseline and after use of alpha lipoic acid. the score range from 0 (worst) to 10 (best)
Vibration Perception Threshold (VPT) | : through study completion, an average of 3 months
  VPT was evaluated using a 128-Hz tuning fork applied bilaterally at the tip of the great toe. Responses were categorized as abnormal (no perception of vibration),present (examiner perceives vibration <10sec after patient reported disappearance of vibration perception) ,and reduced (examiner perceives vibration >10 seconds after patient reported disappearance of vibration perception).
neuromuscular ultrasound | : through study completion, an average of 3 months
  the cross sectional area of the posterior tibial nerve will be assessed in both sides at baseline and after use of alpha lipoic acid
concentration of Hemoglobin A1c | : through study completion, an average of 3 months
  the participants were divided into two categories that include good glycemic control (HA1c≤7%), poor glycemic control (≥ HA1c 7 %),
serum concentrations of high density lipoproteins-cholesterol (HDL-C) | : through study completion, an average of 3 months
  A low HDL cholesterol level was defined as <1.03 mmol/l( 40 mg/dl) for men and <1.29mmol/L(50 mg/dl) for women
serum concentrations of low density lipoproteins-cholesterol (LDL-C) | : through study completion, an average of 3 months
  a patient of LDL-C equal or more than 3.3mmol/L (129mg/dl) is defined as dyslipidemic.
ankle reflex | : through study completion, an average of 3 months
  ranging from 0 (absent) to 4 (hyperactive with clonus)
Measurement of nerve conduction velocity | : through study completion, an average of 3 months
  sensory and motor conduction velocity are measured in meter/second in common peroneal and posterior tibial nerves on both sides at baseline and after use of alpha lipoic acid
measurement of Compound Muscle Action Potential (CMAP) amplitudes | : through study completion, an average of 3 months
  amplitude is measured in micro or millivolts in common peroneal and posterior tibial nerves on both sides at baseline and after use of alpha lipoic acid
measurement of Compound Muscle Action Potential (CMAP) distal latency | : through study completion, an average of 3 months
  distal latency measured in milliseconds and evaluated in common peroneal and posterior tibial nerves on both sides at baseline and after use of alpha lipoic acid

CONTACTS AND LOCATIONS:
Overall Officials: Amira Mohamady, MD, Principal Investigator — Benha university- Qaluibya- Egypt
Locations (1):
- Benha University Hospital, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No